CLINICAL TRIAL: NCT01214967
Title: Empowering Low Income Mothers With Preterm Infants: a Randomized Controlled Trial
Brief Title: Problem Solving Education and Neonatal Intensive Care Unit (NICU) Mothers
Acronym: Project Solve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Tufts Medical Center (Other)
Responsible Party: Principal Investigator, Michael Silverstein, BMC Attending Physician, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Hood-R03HD058075
Record Dates: First submitted 2010-09-27; First posted 2010-10-05 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2010-10

CONDITIONS: Maternal Depression
Keywords: risk factors for maternal depression

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Problem Solving Education, a psycho-educational intervention
  Interventions: Behavioral: Problem Solving Education
- 2 (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Problem Solving Education — psycho-educational intervention
  Arms: 1

SUMMARY:
Premature infants are born at substantial risk for poor health and developmental outcomes, which commonly include hearing and vision problems, developmental delays, and poor school performance. Premature infants of low-income families face additional social risks known to worsen these outcomes. The Institute of Medicine recognized this important public health problem in its 2006 report, Preterm Birth, which argued for the need to improve the quality of follow-up care for preterm infants discharged from the neonatal intensive care unit (NICU). The underpinning of this proposal is that maternal depression - common among families of premature infants - interferes with adherence to follow-up services, and (both through this mechanism and directly) adversely impacts child health and development. Conversely, alleviating depressive symptoms among these women represents a promising strategy to improve adherence to NICU follow-up services and to improve the outcomes of this vulnerable population.

This project aims to mitigate the adverse effects of maternal depression in this specific high-risk population by testing a theory-based, parent-directed empowerment strategy, called Problem Solving Education (PSE). In the past, similar strategies have been proven effective for improving the mood and functioning of depressed adults, and for improving adherence to medical treatment. However, they have never been tested in the setting of a parent-child relationship or among families of premature infants.

This project involves a clinical trial of PSE among 50 low-income mothers at risk for depression, who have premature infants in two Boston NICUs: Boston Medical Center and Tufts Medical Center. The investigators aim to determine the impact of PSE on maternal depressive symptoms and functioning, and adherence to child health supervision and immunization schedules, vision screening, and early intervention evaluation for babies with suspected developmental delays.

Approximately 100,000 children are born prematurely to low-income families each year. Parent-directed PSE aims to improve outcomes for these children through the prevention and/or attenuation of maternal depressive symptoms, as well as through family activation and promotion of adherence to follow-up care. If successful, PSE could also provide the cornerstone of a more generalizable empowerment strategy for families of children with chronic medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Baby is ≤ 33 weeks gestational age and is expected to survive.
* Baby qualifies to receive WIC
* Mother is comfortable in English or Spanish.

Exclusion Criteria:

* Mother has psychosis
* Mother endorses suicidal ideation
* Custody of baby is uncertain
* Mother is cognitively limited, per judgment of NICU attending physician
* Baby is critically ill, per judgment of NICU attending physician

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Maternal Depressive Symptoms | 6 months

SECONDARY OUTCOMES:
Health Care Supervision Schedule for Children | 6 months
Immunization Schedule for Children | 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Boston Medical Center, Boston, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts